CLINICAL TRIAL: NCT00005825
Title: Trans Retinoic Acid (Vesanoid) With Chemotherapy in Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Raghu Nandan, M.D., Inc (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067837; NANDAN-VES-024; NCI-V00-1587
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2003-07

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Mitomycin; Tretinoin; Vinorelbine

INTERVENTIONS:
Drug: cisplatin
Drug: mitomycin C
Drug: tretinoin
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and duration of response to mitomycin, vinorelbine, and cisplatin plus tretinoin in patients with stage IIIB or IV non-small cell lung cancer.
* Determine the toxicity of this treatment regimen in these patients.
* Determine survival of these patients with this treatment regimen.

OUTLINE: Patients receive tretinoin orally twice daily for 4 days starting days 1 and 8; cisplatin IV over 2 hours and vinorelbine IV on days 1 and 8; and mitomycin IV (courses 1 and 3) on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: At total of 15-46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IIIB or IV non-small cell lung cancer
* Measurable disease
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2 times upper limit of normal (ULN)
* AST and ALT less than 2.5 times ULN (unless attributed to liver metastases)

Renal:

* Creatinine no greater than 1.5 mg/dL AND/OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No myocardial infarction within past 6 months
* No congestive heart failure
* No uncontrolled arrhythmia

Other:

* No other concurrent or prior malignancy within past 5 years except localized basal cell or squamous cell skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy with clearly progressive disease
* Concurrent palliative radiotherapy allowed if no evidence of disease progression

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09

CONTACTS AND LOCATIONS:
Overall Officials: Raghu Nandan, MD, Study Chair — Raghu Nandan, M.D., Inc
Locations (1):
- Rajendra Prasad M.D., Inc., Lakewood, California, United States